CLINICAL TRIAL: NCT07258420
Title: The Effect of Using Virtual Reality Glasses on Patients' Anxiety and Comfort Levels in Open Inguinal Hernia Surgery Performed With Spinal Anesthesia
Brief Title: Effect of Watching Video With Virtual Reality Glasses During Surgery on Anxiety and Comfort Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Assos Prof, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-PO189
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Intraoperative; Anxiety; Comfort
Keywords: comfort; nursing care; virtual reality; surgery anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study will be conducted using randomized controlled, experimental type and single blind research methods. For this purpose, after the data is collected, it will be coded as A and B groups, so the researcher who will make the research statistics will analyze the data without knowing the study and control groups. The randomization method will be used to determine the groups. For this, patients who meet the study criteria and volunteer will be assigned to the groups according to the order of their surgery using the 'Random Allocation Software 2.0' randomization program.
Who Masked: Outcomes Assessor
Masking Description: The data analyse is going to be completed by a independent researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will be visited in the rest room in the operating room before the surgery and will be informed about the virtual reality glasses they will use during the surgery. Patients will be asked to watch videos with virtual reality glasses during the surgery. Visual Analog Scale-A was used to assess the anxiety levels of patients and Perioperative Comfort Scale was used to assess their comfort levels
  Interventions: Other: Using a virtual reality glasses
- Control group (No Intervention): Patients in this group will be visited by the researcher in the pre-anesthesia listening room in the operating room before surgery. No other intervention will be made to the patients during surgery. Patients will be visited again in the post-anesthesia recovery room after surgery. Visual Analog Scale-A was used to assess the anxiety levels of the patients; Perioperative Comfort Scale was used to assess their comfort levels.

INTERVENTIONS:
Other: Using a virtual reality glasses — Virtual reality glasses were used on the patients in the study group within the scope of the study. G04EA VR Shinecon 3D Virtual Reality Glasses are compatible with 4.0-6.53 inch Android and IOS smart phones. 3D stereo sound unit is with Bluetooth stereo headset. Due to the use of specially designed resin lenses, it will not cause dizziness or visual fatigue even if worn for a long time. It has IMAX giant screen technology with 720° panoramic view. Flexible, adjustable headband is suitable for most head sizes. Adjustable viewing distance provides maximum comfort.
  Arms: Intervention group

SUMMARY:
This study was conducted to evaluate the effect of using virtual reality glasses during surgery on patients' anxiety and comfort levels. The main hypotheses are as follows:

H1: 'During open inguinal hernia surgery performed with spinal anesthesia, anxiety levels of patients using virtual reality glasses are lower than those of patients who do not use them.' H2: It was determined that 'The comfort levels of patients who use virtual reality glasses during open inguinal hernia surgery performed with spinal anesthesia are higher than those of patients who do not use them'.

Participants will be asked to watch a video using VR goggles during surgery. If there is a comparison group: Researchers will compare patients to a control group to see if there are any differences in anxiety and comfort levels.

DETAILED DESCRIPTION:
Randomization method will be used to determine the groups. Randomization of the patients was done using 'Random Allocation Software 2.0' program and they were divided into 2 groups: 1) Control group and 2) Intervention group.

1. Control Group: Patients in this group will be visited by the researcher in the pre-anesthesia listening room in the operating room before surgery. No other intervention will be made to the patients during surgery. Patients will be visited again in the post-anesthesia recovery room after surgery. Visual Analog Scale-A was used to assess the anxiety levels of the patients; Perioperative Comfort Scale was used to assess their comfort levels.
2. Intervention Group: Patients in this group will be visited by the researcher in the pre-anesthesia recovery room in the operating room before surgery. Patients will be informed about the virtual reality glasses they will use during surgery. Patients will be asked to watch videos with virtual reality glasses during surgery. Patients will be visited again in the post-anesthesia recovery room after surgery. Visual Analog Scale-A was used to assess patients' anxiety levels; Perioperative Comfort Scale was used to assess their comfort levels.

ELIGIBILITY:
Inclusion Criteria:

To research;

* Planned elective surgery
* Those who will undergo inguinal hernia surgery for the first time
* Those who do not have vision, hearing and perception problems
* Patients who want to participate in the study voluntarily were included.

Exclusion Criteria:

* Any anesthesia method other than spinal anesthesia was applied during the procedure
* Under the age of 18, over the age of 75
* Having advanced vision and hearing problems
* Diagnosed with mental and psychological illness
* Using anti-depressant/sedative medication
* Having stopped watching videos during the surgical procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
anxiety level | 18 mounth
  The anxiety levels of the patients will be evaluated with the Visual Analog Scale. It is a measurement tool that can be repeated and requires minimal tools, and is a one-dimensional scale frequently used in the measurement of subjective parameters. VAS is used to convert some values that cannot be measured numerically into numerical values. A 100 mm line is scaled with 10 mm intervals, the two end definitions of the parameter to be evaluated are written on both ends of the line, and the patient is asked to indicate where his/her own situation fits on this line by drawing, putting a dot, or pointing. To evaluate anxiety; "I have no anxiety" labels are placed on the zero point on the line divided into 10 cm, and "I feel a lot of anxiety" labels are placed above the 10th cm.

SECONDARY OUTCOMES:
comfort level | 18 mounth
  The comfort level of the patients will be evaluated with the Perianesthesia Comfort Scale. The lowest total score that can be obtained from the scale is 24, and the highest total score is 144. The average value is found by dividing the total score obtained by the number of scale items and the result is expressed in the 1-6 distribution. Low comfort is expressed with one point, high comfort with six points.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Ünver, Assoc. Prof., Principal Investigator — Trakya University; Esra Çevik, BSN, MSC, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No